CLINICAL TRIAL: NCT06979115
Title: Investigation Into the Safety and Efficacy of ICG-Labeled Fluorescence Imaging Technology in Guiding the Resection of Bone and Soft Tissue Tumors
Acronym: ICG-BST
Status: Not yet recruiting | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ICG-BST
Record Dates: First submitted 2025-04-30; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-03

CONDITIONS: Bone Neoplasms; Soft Tissue Neoplasms
Keywords: Soft tissue neoplasms; Bone neoplasms; Indocyanine green; Near-infrared
MeSH Terms: conditions — Bone Neoplasms; Soft Tissue Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICG Fluorescence Group: For patients with bone and soft tissue tumors, indocyanine green (ICG) is administered intravenously preoperatively. A tailored surgical plan is developed based on tumor location, anatomical complexity, histological subtype, and tumor stage. During surgery, a near-infrared (NIR) fluorescence imaging system is utilized for real-time intraoperative imaging and fluorescence-guided verification of tumor margins. Postoperatively, pathological examination of resected specimens is performed, and the positive margin rate is calculated based on histopathological findings.
  Interventions: Drug: Indocyanine green (ICG)

INTERVENTIONS:
Drug: Indocyanine green (ICG) — Indocyanine green (ICG; National Drug Approval No. H20213567, Ruida Pharmaceuticals) is administered intravenously 24 hours preoperatively at a dose of 2 mg/kg. The drug is dissolved in 250 mL of normal saline using a light-protected infusion set and infused at a constant rate over 60 minutes. Alternatively, a 0.5 mg/kg dose may be administered via IV infusion 1-3 hours before surgery.

SUMMARY:
Investigate the application protocol, feasibility, and efficacy of indocyanine green (ICG)-assisted near-infrared (NIR) fluorescence-guided resection in bone and soft tissue tumors. Assess the incidence of adverse events and evaluate the safety of the protocol.

DETAILED DESCRIPTION:
This research focuses on improving surgical outcomes for patients with bone and soft tissue tumors, a challenging area of cancer treatment. Surgeons face a critical dilemma: removing too much tissue can permanently harm a patient's mobility or function, while removing too little risks leaving behind cancer cells, which may lead to recurrence. Current methods rely heavily on the surgeon's experience and real-time visual or tactile feedback during surgery, but these approaches can be subjective and may miss hidden tumor cells. Traditional tools like frozen tissue analysis during surgery are time-consuming, disrupt the operation, and may not provide accurate results, especially for bone tumors, which require complex processing.

To address these challenges, this study explores an innovative imaging technology called near-infrared (NIR) fluorescence guided surgery, which uses a safe, FDA-approved dye called indocyanine green (ICG). ICG is injected into the patient before surgery and glows under special infrared light, helping surgeons "see" cancer cells in real time. This technology has already proven effective in other cancers (e.g., liver, breast, and colorectal tumors) by highlighting hard-to-detect lesions, guiding lymph node removal, and ensuring complete tumor excision. However, its use in bone and soft tissue tumors-a field with unique anatomical and biological complexities-remains understudied.

Key Goals of the Study:

Tumor Visualization: Test how effectively ICG can "light up" bone and soft tissue tumors under NIR imaging, and determine the optimal timing and methods for administering the dye.

Precision Surgery: Evaluate whether NIR-guided surgery helps surgeons achieve cleaner tumor margins (i.e., removing all cancer cells while sparing healthy tissue).

Accuracy Validation: Compare the fluorescent imaging results with post-surgery pathology reports to confirm if the technology reliably predicts tumor presence.

Practical Insights: Identify factors that might affect the stability and reliability of the imaging system in real-world surgical settings.

Why This Matters:

For Patients: This technology could reduce the risk of cancer recurrence, minimize unnecessary tissue removal, and improve recovery outcomes.

For Surgeons: It offers an objective, real-time tool to enhance decision-making during complex tumor surgeries.

For Cancer Care: If successful, it could establish new standards for precision in orthopedic oncology and inspire broader applications in other understudied cancers.

Real-World Examples:

In liver cancer surgery, ICG has helped surgeons detect tiny, hidden metastases that standard imaging missed.

For lung metastases from sarcoma, ICG-guided removal of suspicious tissue led to a high rate of confirmed cancer cells in additional samples.

Safety and Accessibility:

ICG is widely used in other medical fields, with a strong safety profile approved by global regulatory agencies. The study builds on existing evidence while addressing gaps specific to bone and soft tissue tumors.

By bridging the gap between advanced imaging technology and the unique needs of orthopedic oncology, this research aims to empower surgeons with better tools and give patients a stronger chance at lasting recovery

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of bone and soft tissue tumors (according to the WHO Classification of Tumours of Soft Tissue and Bone, 4th Edition).
2. Medically fit to undergo surgical treatment based on preoperative evaluation.
3. Absence of cardiovascular, anesthesia-related, or other surgical contraindications.

Exclusion Criteria:

1. Presence of severe or chronic kidney, liver, or pulmonary diseases.
2. Autonomous thyroid nodules or allergy to iodine/shellfish.
3. Deemed unable to tolerate surgery based on preoperative evaluation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 40
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-05-25 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Positive Surgical Margin Rate | Within 4 days post-surgery (upon receipt of final pathology report)
  The proportion of cases with tumor cells detected at the surgical margin during postoperative pathological examination, used to assess the completeness of tumor resection.
Positive Residual Lesion Detection Rate | Within 4 days post-surgery (upon receipt of final pathology report)
  The proportion of intraoperatively detected residual lesions (via fluorescence imaging) confirmed as tumor tissue by pathology, reflecting the accuracy of fluorescence imaging in identifying tumor remnants.
Tumor Fluorescence Staining Rate | During surgery
  The success rate of intraoperative tumor visualization using fluorescence imaging after indocyanine green (ICG) injection, evaluating the effectiveness of fluorescence-guided technology.

SECONDARY OUTCOMES:
Local Progression-Free Survival | From the date of surgery until the date of first documented local progression or death from any cause, whichever occurs first, assessed up to 24 months
  The time from surgery to local tumor recurrence or progression, primarily assessing the efficacy of surgery in delaying recurrence.
2-Year Disease-Free Survival (DFS) Rate | Form surgery to 2 years after surgery
  The proportion of patients without tumor recurrence or death within 2 years post-surgery, reflecting intermediate-term treatment efficacy and overall prognosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Data might still be actively analyzed for follow-up studies, and premature sharing could compromise ongoing work or publications.